CLINICAL TRIAL: NCT00168792
Title: A Phase IIIb - IV, Randomised, Open Label Trial Evaluating the Efficacy and Safety of Tenecteplase Together With Unfractionated Heparin Prior to Early PCI as Compared to Standard Primary PCI in Patients With Acute Myocardial Infarction. ASSENT 4 PCI (Assessment of the Safety and Efficacy of a New Treatment Strategy for Acute Myocardial Infarction.)
Brief Title: A Trial Evaluating the Efficacy and Safety of Tenecteplase Together With Unfractionated Heparin Prior to Early Percutaneous Coronary Intervention (PCI) as Compared to Standard Primary PCI in Patients With Acute Myocardial Infarction (ASSENT 4 PCI)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Genentech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123.12
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase
Procedure: PCI

SUMMARY:
To show whether addition of thrombolytic treatment by a single bolus injection of tenecteplase prior to early standard PCI (percutaneous coronary intervention) will improve the clinical outcome in patients with large acute myocardial infarcts as compared to primary PCI alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients giving informed consent
* Patients with a large acute myocardial infarction randomised within 6 hours of symptom onset
* Patients scheduled to undergo primary PCI
* Patients reaching the cath lab not before 60 min and not later than 3 hours after randomisation

(Otherwise the patients fulfill the usual selection criteria for thrombolytic treatment and PCI)

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1671
Dates: Start 2003-11; Primary Completion 2006-07

PRIMARY OUTCOMES:
Death or cardiogenic shock or congestive heart failure within 90 days | 90 days

SECONDARY OUTCOMES:
Death or cardiogenic shock or congestive heart failure within 30 days | 30 days
Cardiogenic shock or congestive heart failure within 90 days | 90 days
Death | 90 days
Cardiogenic shock | 90 days
Reinfarction | 90 days
Repeat target vessel revascularisation (TVR) | 90 days
Rehospitalisation for congestive heart failure | 90 days
Rehospitalisation for cardiogenic shock | 90 days
Rehospitalisation for other cardiac reasons | 90 days
Congestive heart failure | 90 days
N-terminal pro-brain natriuretic peptide (NT pro-BNP) | 90 days
Disabling stroke | 90 days
Total stroke | 90 days
Rehospitalisation for stroke or ICH (intrancranial haemorrhage) | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (176):
- United States (8):
  - Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - Boehringer Ingelheim Investigational Site, Tampa, Florida
  - Boehringer Ingelheim Investigational Site, Macan, Georgia
  - Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - Boehringer Ingelheim Investigational Site, Providence, Rhode Island
- Austria (4):
  - Boehringer Ingelheim Investigational Site, Feldkirch
  - Boehringer Ingelheim Investigational Site, Sankt Pölten
  - Boehringer Ingelheim Investigational Site, Vienna
  - Boehringer Ingelheim Investigational Site, Wiener Neustadt
- Belgium (18):
  - Boehringer Ingelheim Investigational Site, Aalst
  - Boehringer Ingelheim Investigational Site, Anderlecht
  - Boehringer Ingelheim Investigational Site, Angleur
  - Boehringer Ingelheim Investigational Site, Antwerp
  - Boehringer Ingelheim Investigational Site, Bonheiden
  - Boehringer Ingelheim Investigational Site, Bouge
  - Boehringer Ingelheim Investigational Site, Bruges
  - Boehringer Ingelheim Investigational Site, Brussels
  - Boehringer Ingelheim Investigational Site, Charleroi
  - Boehringer Ingelheim Investigational Site, Genk
  - Boehringer Ingelheim Investigational Site, Ghent
  - Boehringer Ingelheim Investigational Site, Gilly
  - Boehringer Ingelheim Investigational Site, Huy
  - Boehringer Ingelheim Investigational Site, La Louvière
  - Boehringer Ingelheim Investigational Site, Leuven
  - Boehringer Ingelheim Investigational Site, Liège
  - Boehringer Ingelheim Investigational Site, Namur
  - Boehringer Ingelheim Investigational Site, Roeselare
- Brazil (6):
  - Boehringer Ingelheim Investigational Site, Blumenau - SC
  - Boehringer Ingelheim Investigational Site, Curitiba - PR
  - Boehringer Ingelheim Investigational Site, Marília - SP
  - Boehringer Ingelheim Investigational Site, Passo Fundo - RS
  - Boehringer Ingelheim Investigational Site, Porto Alegre - RS
  - Boehringer Ingelheim Investigational Site, São Paulo - SP
- Canada (6):
  - Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - Boehringer Ingelheim Investigational Site, Saint-Foy, Ontario
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Regina, Saskatchewan
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Czechia (3):
  - Boehringer Ingelheim Investigational Site, Pardubice
  - Boehringer Ingelheim Investigational Site, Prague
  - Boehringer Ingelheim Investigational Site, Prague 4-Krc
- France (22):
  - Boehringer Ingelheim Investigational Site, Aulnay-sous-Bois
  - Boehringer Ingelheim Investigational Site, Brest
  - Boehringer Ingelheim Investigational Site, Caen
  - Boehringer Ingelheim Investigational Site, Châteauroux
  - Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - Boehringer Ingelheim Investigational Site, Colmar
  - Boehringer Ingelheim Investigational Site, Créteil
  - Boehringer Ingelheim Investigational Site, Lille
  - Boehringer Ingelheim Investigational Site, Lorient
  - Boehringer Ingelheim Investigational Site, Lyon
  - Boehringer Ingelheim Investigational Site, Marseille
  - Boehringer Ingelheim Investigational Site, Massy
  - Boehringer Ingelheim Investigational Site, Metz
  - Boehringer Ingelheim Investigational Site, Montfermeil
  - Boehringer Ingelheim Investigational Site, Montpellier
  - Boehringer Ingelheim Investigational Site, Nice
  - Boehringer Ingelheim Investigational Site, Nîmes
  - Boehringer Ingelheim Investigational Site, Paris
  - Boehringer Ingelheim Investigational Site, Perpignan
  - Boehringer Ingelheim Investigational Site, Pontoise
  - Boehringer Ingelheim Investigational Site, Saint-Etienne
  - Boehringer Ingelheim Investigational Site, Strasbourg
- Germany (37):
  - Boehringer Ingelheim Investigational Site, Bad Friedrichshall
  - Boehringer Ingelheim Investigational Site, Bad Kreuznach
  - Boehringer Ingelheim Investigational Site, Bassum
  - Boehringer Ingelheim Investigational Site, Bautzen
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Bingen
  - Boehringer Ingelheim Investigational Site, Bonn
  - Boehringer Ingelheim Investigational Site, Boppard
  - Boehringer Ingelheim Investigational Site, Böblingen
  - Boehringer Ingelheim Investigational Site, Bremen
  - Boehringer Ingelheim Investigational Site, Cologne
  - Boehringer Ingelheim Investigational Site, Dresden
  - Boehringer Ingelheim Investigational Site, Fürstenfeldbruck
  - Boehringer Ingelheim Investigational Site, Gransee
  - Boehringer Ingelheim Investigational Site, Hamelin
  - Boehringer Ingelheim Investigational Site, Heidelberg
  - Boehringer Ingelheim Investigational Site, Jena
  - Boehringer Ingelheim Investigational Site, Kassel
  - Boehringer Ingelheim Investigational Site, Kiel
  - Boehringer Ingelheim Investigational Site, Koblenz
  - Boehringer Ingelheim Investigational Site, Korbach
  - Boehringer Ingelheim Investigational Site, Leipzig
  - Boehringer Ingelheim Investigational Site, Lichtenberg
  - Boehringer Ingelheim Investigational Site, Ludwigsburg
  - Boehringer Ingelheim Investigational Site, Mannheim
  - Boehringer Ingelheim Investigational Site, Minden
  - Boehringer Ingelheim Investigational Site, Möckmühl
  - Boehringer Ingelheim Investigational Site, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Offenbach
  - Boehringer Ingelheim Investigational Site, Öhringen
  - Boehringer Ingelheim Investigational Site, Paderborn
  - Boehringer Ingelheim Investigational Site, Ravensburg
  - Boehringer Ingelheim Investigational Site, Rüdesheim am Rhein
  - Boehringer Ingelheim Investigational Site, Schwalmstadt
  - Boehringer Ingelheim Investigational Site, Sömmerda
  - Boehringer Ingelheim Investigational Site, Wiesbaden
- Greece (7):
  - Boehringer Ingelheim Investigational Site, Athens
  - Boehringer Ingelheim Investigational Site, Heraklion
  - Boehringer Ingelheim Investigational Site, Ioannina
  - Boehringer Ingelheim Investigational Site, Nea Efkarpia/ Thessaloniki
  - Boehringer Ingelheim Investigational Site, Nikaea, Piraeus
  - Boehringer Ingelheim Investigational Site, Rio, Patra
  - Boehringer Ingelheim Investigational Site, Thessaloniki
- Hungary (4):
  - Boehringer Ingelheim Investigational Site, Balatonfüred
  - Boehringer Ingelheim Investigational Site, Budapest
  - Boehringer Ingelheim Investigational Site, Debrecen
  - Boehringer Ingelheim Investigational Site, Pécs
- Boehringer Ingelheim Investigational Site, Galway, Ireland
- Italy (30):
  - Boehringer Ingelheim Investigational Site, Alessandria
  - Boehringer Ingelheim Investigational Site, Bassano del Grappa
  - Boehringer Ingelheim Investigational Site, Caserta
  - Boehringer Ingelheim Investigational Site, Catania
  - Boehringer Ingelheim Investigational Site, Cremona
  - Boehringer Ingelheim Investigational Site, Florence
  - Boehringer Ingelheim Investigational Site, Genova
  - Boehringer Ingelheim Investigational Site, Lecce
  - Boehringer Ingelheim Investigational Site, Lecco
  - Boehringer Ingelheim Investigational Site, Loreto Mare (NA)
  - Boehringer Ingelheim Investigational Site, Mantova
  - Boehringer Ingelheim Investigational Site, Massa
  - Boehringer Ingelheim Investigational Site, Messina
  - Boehringer Ingelheim Investigational Site, Mirano (VE)
  - Boehringer Ingelheim Investigational Site, Monza
  - Boehringer Ingelheim Investigational Site, Novara
  - Boehringer Ingelheim Investigational Site, Padua
  - Boehringer Ingelheim Investigational Site, Palermo
  - Boehringer Ingelheim Investigational Site, Pesaro
  - Boehringer Ingelheim Investigational Site, Potenza
  - Boehringer Ingelheim Investigational Site, Ravenna
  - Boehringer Ingelheim Investigational Site, Rho (mi)
  - Boehringer Ingelheim Investigational Site, Roma
  - Boehringer Ingelheim Investigational Site, Salerno
  - Boehringer Ingelheim Investigational Site, San Donato Milanese
  - Boehringer Ingelheim Investigational Site, Sassari
  - Boehringer Ingelheim Investigational Site, Torino
  - Boehringer Ingelheim Investigational Site, Udine
  - Boehringer Ingelheim Investigational Site, Varese
  - Boehringer Ingelheim Investigational Site, Zingonia (bg)
- Mexico (6):
  - Boehringer Ingelheim Investigational Site, Col. Doctores
  - Boehringer Ingelheim Investigational Site, Col. Granada
  - Boehringer Ingelheim Investigational Site, Col. Magdalena de Las Salinas
  - Boehringer Ingelheim Investigational Site, Col. Sección XVI, Deleg.
  - Boehringer Ingelheim Investigational Site, Col. Valle Verde
  - Boehringer Ingelheim Investigational Site, Mèxico, D.F.
- Norway (2):
  - Boehringer Ingelheim Investigational Site, Bergen
  - Boehringer Ingelheim Investigational Site, Oslo
- Poland (10):
  - Boehringer Ingelheim Investigational Site, Katowice
  - Boehringer Ingelheim Investigational Site, Katowice-Ochojec
  - Boehringer Ingelheim Investigational Site, Krakow
  - Boehringer Ingelheim Investigational Site, Lodz
  - Boehringer Ingelheim Investigational Site, Lublin
  - Boehringer Ingelheim Investigational Site, Opole
  - Boehringer Ingelheim Investigational Site, Poznan
  - Boehringer Ingelheim Investigational Site, Warsaw
  - Boehringer Ingelheim Investigational Site, Wroclaw
  - Boehringer Ingelheim Investigational Site, Zabrze
- Portugal (7):
  - Boehringer Ingelheim Investigational Site, Almada
  - Boehringer Ingelheim Investigational Site, Amadora
  - Boehringer Ingelheim Investigational Site, Carnaxide
  - Boehringer Ingelheim Investigational Site, Coimbra
  - Boehringer Ingelheim Investigational Site, Lisbon
  - Boehringer Ingelheim Investigational Site, Porto
  - Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
- Thailand (2):
  - Boehringer Ingelheim Investigational Site, Bangkok
  - Boehringer Ingelheim Investigational Site, Chiang Mai
- Turkey (Türkiye) (3):
  - Boehringer Ingelheim Investigational Site, Ankara
  - Boehringer Ingelheim Investigational Site, Istanbul
  - Boehringer Ingelheim Investigational Site, Izmir

REFERENCES:
- [Result] Assessment of the Safety and Efficacy of a New Treatment Strategy with Percutaneous Coronary Intervention (ASSENT-4 PCI) investigators. Primary versus tenecteplase-facilitated percutaneous coronary intervention in patients with ST-segment elevation acute myocardial infarction (ASSENT-4 PCI): randomised trial. Lancet. 2006 Feb 18;367(9510):569-78. doi: 10.1016/S0140-6736(06)68147-6. PMID 16488800
- [Derived] Zalewski J, Bogaerts K, Desmet W, Sinnaeve P, Berger P, Grines C, Danays T, Armstrong P, Van de Werf F. Intraluminal thrombus in facilitated versus primary percutaneous coronary intervention: an angiographic substudy of the ASSENT-4 PCI (Assessment of the Safety and Efficacy of a New Treatment Strategy with Percutaneous Coronary Intervention) trial. J Am Coll Cardiol. 2011 May 10;57(19):1867-73. doi: 10.1016/j.jacc.2010.10.061. PMID 21545942
- [Derived] Jarai R, Huber K, Bogaerts K, Sinnaeve PR, Ezekowitz J, Ross AM, Zeymer U, Armstrong PW, Van de Werf FJ; ASSENT-4 PCI investigators. Prediction of cardiogenic shock using plasma B-type natriuretic peptide and the N-terminal fragment of its pro-hormone [corrected] concentrations in ST elevation myocardial infarction: an analysis from the ASSENT-4 Percutaneous Coronary Intervention Trial. Crit Care Med. 2010 Sep;38(9):1793-801. doi: 10.1097/CCM.0b013e3181eaaf2a. PMID 20562693